CLINICAL TRIAL: NCT07344129
Title: The Effect of Using the Learning in Pairs (LiP) Model in Episiotomy Education on Students' Episiotomy Knowledge, Self-Efficacy, and Anxiety Levels
Brief Title: Learning in Pairs in Episiotomy Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Şilan YAVUZ, Research Assistant, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 12122025
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Episiotomy; Learning in Pairs
Keywords: episiotomy; learning in pairs; midwifery; self-afficacy; anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The control group will undergo episiotomy in the cow tongue group. The learning group will undergo episiotomy in pairs.
Who Masked: Outcomes Assessor
Masking Description: The control group will undergo episiotomy in the cow tongue group. The learning group will undergo episiotomy in pairs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (application with calf tongue) (No Intervention): At Sakarya University Midwifery Department, episiotomy laboratory practice is routinely performed on calf tongues under instructor supervision as part of the Normal Birth and Postpartum Period course.Therefore, the group performing the practice on calf tongues has been accepted as the control group.The instructor will first provide theoretical training on episiotomy to the group arriving at the laboratory.The training content includes the importance of episiotomy, its risks, indications, contraindications, timing of episiotomy, materials used, types of episiotomy, episiotomy repair and timing, suture techniques, and midwifery care in episiotomy.Immediately after the training, episiotomy repair (suture techniques) will be practiced.Eight students will be accepted for the practice at the same time, and each student will sit at a single-person practice table.The instructor will try to pay attention to each student and will assist with suture techniques as long as the student requests it.
- Experimental group (Application with learning in pairs) (Experimental): The instructor first provides the group arriving at the episiotomy laboratory with theoretical training on episiotomy,covering the importance of episiotomy,its risks, indications, contraindications, timing of episiotomy,materials used,types of episiotomy,episiotomy repair-timing, suture techniques,midwifery care in episiotomy.At the end of the theoretical training,they will watch videos related to suture techniques.After the training, they will proceed to the episiotomy repair(suture techniques) application.Students will be taken to the laboratory in pairs.A maximum of 4 pairs of students will be taken to the laboratory at the same time.The pairs will share the same table.Students will be instructed to begin episiotomy repair on a calf tongue in accordance with their episiotomy application knowledge and skills and to perform the repair procedure by supporting each other during the repair.Students are expected to repair the incision on the calf tongue separately in pairs.
  Interventions: Other: Application with learning in pairs

INTERVENTIONS:
Other: Application with learning in pairs — Students will be taken to the laboratory in pairs. A maximum of 4 pairs of students will be taken to the laboratory at the same time. The pairs will share the same table. Students will be instructed to begin episiotomy repair on a calf tongue in accordance with their episiotomy application knowledge and skills and to perform the repair procedure by supporting each other during the repair. Students are expected to repair the incision on the calf tongue separately in pairs.
  Arms: Experimental group (Application with learning in pairs)

SUMMARY:
There are significant shortcomings in current educational practices regarding midwives acquiring episiotomy skills. The acquisition of episiotomy skills by midwifery students begins in episiotomy skills laboratories. Students acquiring these skills in the laboratory involves being able to assess the indications for episiotomy and perform appropriate interventions based on the indication. Numerous intervention studies have been conducted on teaching episiotomy skills to students. In most of these studies, sponges, chickens, and cow tongues were preferred as simulators, and the effectiveness of the training was evaluated by applying different teaching methods. In addition to simulators used in episiotomy training, there are teaching methods used in midwifery clinical education, one of which is the paired learning model. This study was designed as a randomized controlled trial to evaluate the effect of the learning in pairs model in episiotomy training on episiotomy knowledge level, episiotomy self-efficacy, and state anxiety levels among midwifery students. The study will be conducted with a total of 92 midwifery students, divided into an intervention group (n=46) and a control group (n=46) (1:1 ratio). Data will be collected using the "Student Information Form," "Episiotomy Information Form," "Episiotomy Self-Efficacy Scale," and "State Anxiety Inventory" in pre-test and post-test formats. The research sample will consist of all students enrolled in the midwifery program and the Normal Birth and Postpartum Period course who agree to participate in the study. At the end of the study, it is expected that the effects of the learning in pairs (LiP) model on students' learning in episiotomy repair training will be explained. It is believed that the research results will contribute to midwifery education by enriching the methods used in midwifery students' education.

DETAILED DESCRIPTION:
Childbirth is a significant turning point in a woman's life and can occur either spontaneously or with intervention. In assisted births, episiotomy and its repair are among the most commonly performed interventions, and midwives play an active role in episiotomy repair. Episiotomy is a common surgical incision made in the bulbocavernosus muscle at the end of the second stage of labor to reduce the risk of laceration and preserve perineal tone (Ahmed et al., 2023; Ghulmiyyah et al., 2022). A study conducted with midwifery students reported a deficiency in the current educational practices of midwives regarding episiotomy (Webb et al., 2021). In particular, a lack of confidence was observed in the decision-making mechanisms regarding when and how to perform clinically indicated episiotomies, especially in recognizing the indications for episiotomy (Gould et al., 2023). There are significant deficiencies in current educational practices regarding midwives' acquisition of episiotomy skills (Webb et al., 2021). Teaching episiotomy skills to midwifery students begins in episiotomy skills laboratories. Students acquiring these skills in the laboratory involves being able to assess the indications for episiotomy and perform the appropriate interventions based on the indication. However, being monitored and observed by the instructor during skills training can cause anxiety in students. The anxiety felt by students can negatively affect the learning process, reducing their success levels and self-efficacy (Demirel et al., 2020). Many intervention studies have been conducted on the type of intervention, anxiety, and self-efficacy levels in teaching episiotomy skills to students. In most of these studies, sponge, chicken, and calf tongue were preferred as simulators, and the effectiveness was evaluated by applying different teaching methods (Gönenç et al., 2025; Yılar Erkek & Öztürk Altınayak, 2021; Yolcu et al., 2025). In a study using a calf tongue model, participants reported that this model was similar to perineal injury repair in clinical practice (Faithfull-Byrne et al., 2017). In a study using a chicken model, it was determined that it was an effective educational material in increasing midwifery students' perceived confidence in performing episiotomy, but no significant difference was found in terms of its effect on their anxiety levels (Gönenç et al., 2025). In a systematic review evaluating the effectiveness of simulation methods used in episiotomy training, studies using a calf tongue simulator reported that students had higher self-confidence scores compared to those using a sponge model. In a study using only the calf tongue, it was observed that the calf tongue reduced students' anxiety levels and increased their self-efficacy levels (Şen Aytekin et al., 2022). Self-efficacy is an important factor in the process of students acquiring skills, and in every application, the acquired skill should be measured concretely and the level of contribution of the application to education should be proven (Demirel et al., 2020).

One of the methods used in midwifery clinical education is the learning in pairs (LiP) model. The learning in pairs model offers collaborative learning opportunities in clinical practice, making it a beneficial and alternative approach to clinical learning, especially when mentors are insufficient (Hill et al., 2020; Widarsson et al., 2025). In this approach, students are guided and supported to work collaboratively with other students under the guidance of a coach to provide patient- or practice-focused care. The coach is a mentor who works with groups of 3-6 students in their field, using only coaching approaches in student supervision. The coach encourages students and, rather than providing them with answers, communicates with them and draws on their knowledge. Student groups receive coaching to provide care in a placement setting (clinic, laboratory, etc.) and to work with other students. In the peer learning model, coaching is a fundamental feature of the learning philosophy. The student's knowledge, questioning power in guidance, ability to collaborate, and taking responsibility are other fundamental characteristics of this model (Faithfull-Byrne et al., 2017; Hill et al., 2020). To the best of our knowledge, there is no literature on a study where this model, primarily applied in the clinic, has been implemented with midwifery students in episiotomy laboratories-which can be considered the preclinical setting of midwifery clinics-using simulators. Therefore, this study aimed to evaluate the effect of episiotomy application training given with the calf tongue and paired learning model on midwifery students' episiotomy knowledge level, episiotomy self-efficacy, and state anxiety levels.

ELIGIBILITY:
Inclusion Criteria:

* Students who agree to participate in the study,
* Students enrolled in the midwifery program,
* Students enrolled in the Normal Birth and Postpartum Period course.

Exclusion Criteria:

* Students who did not attend the theoretical part of the episiotomy course,
* Students who did not attend the episiotomy laboratory course,
* Students who have previously taken the Normal Birth and Postpartum Period course and have experience in episiotomy skills.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2026-01-09 (Estimated); Study Completion 2026-01-16 (Estimated)

PRIMARY OUTCOMES:
State Anxiety Inventory (STAI) | 2 hours
  The inventory consists of a total of 20 items. Ten items (items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20) in the state anxiety section are reverse-coded. The inventory is a 4-point Likert scale rated as "Not at all," "A little," "A lot," and "Completely." The total weighted score obtained for direct statements is calculated by subtracting the total weighted score of reverse statements and adding a fixed value (35 points) to this number. The total score ranges from 20 to 80. A high score on the inventory indicates a high level of anxiety, while a low score indicates a low level of anxiety.
Episiotomy Self-Efficacy Scale | 2 hours
  The scale consists of a total of 17 items and four subscales (cognitive, emotional, motivational, and psychomotor). The scale is a 5-point Likert scale, and the ratings are (1) Strongly Disagree, (2) Somewhat Disagree, (3) Undecided, (4) Somewhat Agree, (5) Strongly Agree. There are no reverse-coded items on the scale. The lowest possible total score on the scale is 17, and the highest possible score is 85. High scores on the scale indicate high episiotomy self-efficacy. The Cronbach's Alpha reliability coefficient for the scale as a whole is reported as 0.955.
Episiotomy Information Form | 2 hours
  This form consists of 25 statements (questions) designed to measure students' level of knowledge about episiotomy. Thirteen of these statements are true, and twelve are false. Participants are asked to respond with "True," "False," or "I don't know." Students' "True" responses to the statements will be scored as 1 point, while 'False' and "No opinion" responses will be scored as 0 points. The lowest possible score on the knowledge form is 0, and the highest possible score is 25.

REFERENCES:
- [Background] Yolcu B, Kaymak ZD, Turan Z, Baskaya YH. The episiotomy self-efficacy scale: a scale development study. BMC Nurs. 2025 Jul 17;24(1):931. doi: 10.1186/s12912-025-03578-9. PMID 40676655
- [Background] Yılar Erkek, Z., & Öztürk Altınayak, S. (2021). The Effect of Simulation Teaching Technique on the Improvement of Episiotomy Performance Skills and State Anxiety of Midwifery Students in Turkey: RCT. Clinical Simulation in Nursing, 54, 62-69. https://doi.org/10.1016/j.ecns.2021.01.014
- [Background] Widarsson M, Velandia M, Pellfolk MG, Kerstis B. Learning in pairs in Swedish delivery wards: A win-win approach for midwifery preceptors and students. Midwifery. 2025 Dec;151:104632. doi: 10.1016/j.midw.2025.104632. Epub 2025 Oct 11. PMID 41124872
- [Background] Webb SS, Skene ER, Manresa M, Percy EK, Freeman RM, Tincello DG. Evaluation of midwifery pelvic floor education and Training across the UK and Spain. Eur J Obstet Gynecol Reprod Biol. 2021 Jan;256:140-144. doi: 10.1016/j.ejogrb.2020.10.065. Epub 2020 Nov 5. PMID 33227686
- [Background] Spielberger, C. D., Gorsuch, R. L., Lushene, R., Vagg, P., & Jacobs, G. (1983). State-Trait Anxiety Inventory For Adults . Consulting Psychologists Press, Palo Alto, CA.
- [Background] Şen Aytekin, M., Kahraman, A., & Alparslan, Ö. (2022). Ebelik Öğrencilerine Epizyotomi Öğretmeye Yönelik Kullanılan Simülasyon Yöntemlerinin Etkisi: Sistematik Derleme. J TOGU Heal Sci, 2(2), 212-224.
- [Background] Öner, N., & Le Compte, A. (1983). State-trait anxiety inventory handbook. Boğaziçi University Publications, 333, 1-26.
- [Background] Hill R, Woodward M, Arthur A. Collaborative Learning in Practice (CLIP): Evaluation of a new approach to clinical learning. Nurse Educ Today. 2020 Feb;85:104295. doi: 10.1016/j.nedt.2019.104295. Epub 2019 Nov 21. PMID 31783268
- [Background] Gould J, Webb SS, Byrne C, Brace E, Cleary J, Dow L, Edwards E, Glyn-Jones E, Hunter T, Longton J, Tibble K, MacLellan J. Red flags for episiotomy in a midwife-led birth: Using co-production with midwives to capture clinical experience. Women Birth. 2023 Mar;36(2):217-223. doi: 10.1016/j.wombi.2022.06.009. Epub 2022 Aug 6. PMID 35941059
- [Background] Gönenç, İ. M., Aker, M. N., & Alan Dikmen, H. (2025). The Effect of Chicken Model on Satisfaction, Self-Confidence, and Anxiety in Teaching Episiotomy Repair: A Randomized Controlled Trial. Turkiye Klinikleri Journal of Health Sciences, 10(3), 647-657. https://doi.org/10.5336/healthsci.2025-108536
- [Background] Ghulmiyyah L, Sinno S, Mirza F, Finianos E, Nassar AH. Episiotomy: history, present and future - a review. J Matern Fetal Neonatal Med. 2022 Apr;35(7):1386-1391. doi: 10.1080/14767058.2020.1755647. Epub 2020 Apr 26. PMID 32338105
- [Background] Faithfull-Byrne, A., Thompson, L., Schafer, K. W., Elks, M., Jaspers, J., Welch, A., Williamson, M., Cross, W., & Moss, C. (2017). Clinical coaches in nursing and midwifery practice: Facilitating point of care workplace learning and development. Collegian, 24(4), 403-410. https://doi.org/10.1016/j.colegn.2016.06.001
- [Background] Demirel, G., Evcili, F., Kaya, N., & Doganer, A. (2020). The Effect of Episiotomy Repair Simulation on the Anxiety and Self-Efficacy levels of Midwifery Students. Journal of Midwifery and Reproductive Health, 8(1), 2050-2057. https://doi.org/10.22038/jmrh.2019.42024.1479
- [Background] Ahmed M, Kaur I, Thota S. Changing minds: The impact of introducing evidence-based practices around the use of episiotomy in a South Indian Tertiary Centre. Midwifery. 2023 Nov;126:103833. doi: 10.1016/j.midw.2023.103833. Epub 2023 Sep 25. PMID 37801839